CLINICAL TRIAL: NCT01351142
Title: Cytokines and Cognitive Decline in Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Allocation: Not Applicable | Model: Single Group
Other Study IDs: CYTOCOGMA
Record Dates: First submitted 2011-05-06; First posted 2011-05-10 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Hematologic Tests; Neuropsychological Tests

INTERVENTIONS:
Other: blood test and cognitive tests — Specific cognitive tests are performed at day 1, month 6, one year and 2 years Specific Blood samples tests are performed at inclusion, 1 years and 2 years

SUMMARY:
Amyloid plaques and neurofibrillary tangles are the 2 well-known etiopathological hallmarks of Alzheimer's disease (AD). Beside these 2 lesions, inflammation response is described in the brain of patients with AD.

The main objective of our study is to analyse the correlation between the value of plasma cytokines (interleukin 1, 6, TNFα and chemochine Rantes) and the rapidity of the cognitive decline in AD over a 2-year follow-up.

Secondary objectives include:

* the predictive value of the cytokines on the cognitive decline after 6 months and one year of follow-up., of the patients include 150 patients with AD (MMSE: 16-25)
* correlation between plasma cytokines levels and expression of the protein kinase PKR (involved in death cell) in blood mononuclear cells.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease (AD)patients
* MMSE score: 16-25
* Written informed consent

Exclusion Criteria:

* AD patients with specific treatment for AD before inclusion MMSE score under 16 or over 25 at inclusion
* patients with anti-inflammatory drugs (non steroids or corticosteroids) or immunosuppressive agents
* Patients with acute disease (infectious disease, rheumatologic disease) or chronic disease (malignancy, infectious, rheumatologic disease) that could interact with plasma cytokines level
* Patients with a life threatening disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2009-11; Primary Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU Angers - service Gérontologie clinique, Angers
  - Hôpital Dupuytren - CHU de Limoges, Limoges
  - CHU de NANTES - service Gériatrie, Nantes
  - CHU DE NANTES - Centre ambulatoire de Gérontologie clinique, Nantes
  - Hôpital Broca - service de Gériatrie, Paris
  - Hôpital Pitié Salpétrière, Paris
  - Chu de Poitiers -, Poitiers
  - Chu Strasbourg, Strasbourg
  - CHU de TOURS - service de Gériatrie, Tours
  - Hôpital gériatrique des Charpennes, Villeurbanne